CLINICAL TRIAL: NCT00361478
Title: Effect of the 'Mother and Baby' Program on New Mothers' Psychological and Physical Well-Being.
Brief Title: Effect of the 'Mother and Baby' Program on Well-Being
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Dr Mary Galea, The University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07/2004
Record Dates: First submitted 2006-08-07; First posted 2006-08-08 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2006-07

CONDITIONS: Postnatal Depression
Keywords: exercise; postnatal depression; psychological health; well-being
MeSH Terms: conditions — Depression, Postpartum; Motor Activity; Psychological Well-Being | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): "Mother and Baby" Program comprising exercise and education.
  Interventions: Behavioral: Exercise and education
- 2 (Active Comparator): Education only
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Exercise and education — Weekly exercise and education program for 8 weeks
  Other Names: Exercise
  Arms: 1
Behavioral: Education — Written educational material
  Other Names: Educational material
  Arms: 2

SUMMARY:
The study investigates the effect of the 'Mother and Baby' (M&B) program on the psychological health and well-being of new mothers 6-10 weeks following the birth of their baby. The M&B program is an 8-week program of group exercise and education sessions provided by various health professionals. The design of the study is a comprehensive cohort design, including a randomised controlled trial. The primary outcome measure is the Affect Balance Scale. The hypotheses are:

1. The M&B program has a positive effect on new mothers' psychological health and well-being.
2. The M&B program increases participation in regular physical activity.
3. the M&B program benefits first time mothers more than women who have had more than one child.

DETAILED DESCRIPTION:
Background

The benefits of exercise, in particular group exercise, for women in early motherhood include improved body image, decreased anxiety, improved energy and building of social networks. Exercise has also been shown to be beneficial in the management of mood disorders such as depression and more specifically, postnatal depression. However there has been no suggestion that exercise may reduce symptoms of psychotic disorders that require medication, psychiatric therapy and possible hospitalisation. The number of women experiencing postnatal depression (PND) has increased to one in five women following childbirth. Some of the risks of development of PND include lack of social support during the childbearing year and lack of involvement in the community. new mothers have identified that reasons for inactivity include no child care, limited opportunity to exercise with their baby, reduced self-esteem, poor body image, or they are too busy. Research to date is limited and qualitative in nature, with no standardised measurement tools used to assess quality of life in postnatal women.

The 'Mother and Baby' (M&B) program is an 8-week program involving one hour of group exercise with mothers and their babies conducted by a physiotherapist and a 30-minute education session provided by various health professionals (physiotherapist, nutritionist, speech pathologist, psychologists and midwives). Education topics include baby massage, nutrition for mothers, introducing solids, adjusting to a new lifestyle, communicating with the baby, sun care for the baby and play development. The aim of the study is to explore the benefits of the M&B program on new mothers' psychological and physical well-being as well as the social benefits of exercise.

Research Plan

The design of the study is a comprehensive cohort design incorporating a randomised controlled trial (RCT)of the effects of the M&B program on the health of health women 6-10 weeks following the birth of their baby. The cohort design will complement the results of a classic RCT by allowing the investigation of outcomes in a setting that simulates the 'real-world' treatment process.

Women who have had their babies at the Angliss Hospital and are ready for discharge will be invited to participate in the study. Potential participants will be asked if they have a preference for the M&B program or Education sessions only, or if they would be willing to be part of an RCT. Those who agree to be part of the RCT will be randomised to M&B or Education only sessions. Allocation will be controlled by the chief investigator and will be concealed, with codes placed in opaque sealed enveloped. Randomisation will be stratified according to parity (first time mothers vs multiparous) and blocked in groups of 16.

All participants will receive and complete a questionnaire booklet and will return this in a pre-paid envelope. Questionnaires include:

1. The Affect Balance Scale. This is the primary outcome measure. It is a highly reliable scale comprising ten questions indicating psychological reactions (positive and negative) to events in daily life.
2. Edinburgh Postnatal Depression Scale. This is a widely used scale for the detection of risk factors for postnatal depression.
3. Questions regarding exercise. Three questions regarding exercise will be asked and answers will be compared to tables of the number of metabolic equivalents (METS) required to perform the activity.
4. Program evaluation. Participants undertaking the M&B program will complete a standardised evaluation form.

Sample size

A preliminary power calculation has been conducted from studies using the Affect Balance Scale in similar settings. With 80 subjects per group we will have 80% power to detect a 1.4 unit difference between the two groups. An advantage of 1.4 units (or 7% to 10% across a scale) is regarded as a clinically important difference. A pilot study will be undertaken to confirm the sample size.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women giving birth at the Angliss Hospital (primiparous and multiparous)

Exclusion Criteria:

* Previous history of postnatal depression

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2005-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Affect Balance Scale | 4 weeks

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale | 4 weeks
Exercise level | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Galea, PhD, Study Director — University of Melbourne; Emily Ashby, BPhysio, Principal Investigator — The Angliss Hospital; Margaret Sherburn, MWHlth, Principal Investigator — University of Melbourne; Richard Osborne, PhD, Principal Investigator — University of Melbourne
Locations (1):
- The Angliss Hospital, Ferntree Gully, Victoria, Australia

REFERENCES:
- [Derived] Norman E, Sherburn M, Osborne RH, Galea MP. An exercise and education program improves well-being of new mothers: a randomized controlled trial. Phys Ther. 2010 Mar;90(3):348-55. doi: 10.2522/ptj.20090139. Epub 2010 Jan 7. PMID 20056720